CLINICAL TRIAL: NCT04442802
Title: Rate of Severe Arterial Dissections After Femoropopliteal Angioplasty by Long Versus Short Time of Balloon Inflation: the LOVES Randomized Controlled Trial
Brief Title: Arterial Dissections After Angioplasty by Long vs Short Time of Balloon Inflation: the Randomized Controlled Trial.
Acronym: LOVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dumitru Casian (Other)
Responsible Party: Sponsor-Investigator, Dumitru Casian, Associate Professor Department of General surgery nr.3, Head of Vascular Surgery Clinic, Universitatea de Stat de Medicina si Farmacie Nicolae Testemiţanu
Organization: Universitatea de Stat de Medicina si Farmacie Nicolae Testemiţanu (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOVES_RCT_2020
Record Dates: First submitted 2020-06-16; First posted 2020-06-23 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease; Dissection Arterial
MeSH Terms: conditions — Peripheral Arterial Disease; Aortic Dissection | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long time balloon inflation (Experimental): During the endovascular intervention the angioplasty balloon will be inflated for 6 minutes to treat the occlusive-stenotic femoropopliteal arterial lesion
  Interventions: Procedure: Percutaneous transluminal angioplasty
- Short time balloon inflation (Active Comparator): During the endovascular intervention the angioplasty balloon will be inflated for 3 minutes to treat the occlusive-stenotic femoropopliteal arterial lesion
  Interventions: Procedure: Percutaneous transluminal angioplasty

INTERVENTIONS:
Procedure: Percutaneous transluminal angioplasty — Under local anesthesia the percutaneous arterial access will be created. Digital subtraction angiography of the whole limb will be performed. Occlusive-stenotic lesion of the superficial femoral and / or popliteal artery will be crossed with a guidewire. The plain old (non drug-eluting) will be positioned in the affected arterial segment and inflated up to nominal pressure. After balloon deflation and extraction the completion angiography will be performed. Presence (yes/no) and severity (grades A-B or C-F according to NHLBI classification) of dissection will be assessed independently by 3 study investigators basing on DSA images in 2 directions. Decision to classify the dissection as severe (grade C-F) and to perform the bailout stenting will be done by the agreement between at least 2 from 3 investigators.
  Other Names: Plain old balloon angioplasty

SUMMARY:
Background. Arterial dissections represent the typical complication of the percutaneous transluminal angioplasty for femoropopliteal disease and have negative impact upon the outcomes of the treatment.

Objective. The study is aimed to test the hypothesis that a prolonged (6 minutes) time of inflation of angioplasty balloon would reduce the rate of severe arterial dissections and necessity in bailout stenting during the treatment of occlusive-stenotic femoropopliteal lesions in patients with chronic limb threatening ischemia.

Methods. The LOVES trial is a single centre, two parallel groups, controlled trial with 1:1 randomization. Participants will be recruited among the patients hospitalized in Vascular Surgery Department of Institute of Emergency Medicine, Chisinau, Republic of Moldova.

Procedure. Diagnostic angiography of the treated limb will be performed first to confirm the presence of stenosis ≥50% or occlusion in the superficial femoral and/or popliteal artery. After crossing of the lesion patient will be supposed to randomization. In the intervention group the angioplasty balloon will be inflated for 6 minutes. In the control group - for 3 minutes.

Presence and severity (grades A-B or C-F according to NHLBI classification) of dissection will be assessed independently by 3 study investigators basing on completion angiography. Decision to classify the dissection as severe (grade C-F) and to perform the bailout stenting will be done by the agreement between at least 2 investigators.

Sample size. Basing on the results of previous retrospective study investigators expect the 23% rate of severe dissection in study group (6 minutes inflation) and 51% - in control group (3 minutes inflation). Using the probability of type I error of 0.05 and power set at 80% investigators have calculated that 45 patients are required for each group. Anticipating 10% rate of loss to follow-up, 50 patients will be randomized per treatment arm.

Randomization. One hundred patients will be allocated to study or control group by two blocks 1:1 randomization using the free online application Research Randomizer, version 4 (Urbaniak GC, Plous S., 2013, http://www.randomizer.org/).

Follow-up. Three follow up visits at 1, 6 and 12 months are scheduled.

DETAILED DESCRIPTION:
Background. Arterial dissections represent the typical complication of the percutaneous transluminal angioplasty for femoropopliteal disease, with an incidence of 20-60% depending of the severity of treated lesion and reporting standards. Post-angioplasty dissections have negative impact upon the outcomes of the endovascular treatment of lower limb arterial disease. Severe flow limiting dissections require immediate treatment by bailout stenting. Although this strategy is effective in the short term there is a substantial risk of in-stent restenosis, stent thrombosis, and stent fracture with the long-term follow-up. Moreover, it was demonstrated that even minor dissections that required no treatment during the initial procedure with time can progress to significant arterial stensosis. Finally, stenting significantly increases the cost of intervention.

Improved results of peripheral arterial balloon angioplasty with balloon inflation time of 3 minutes comparing to 1 minute were reported previously. A randomized study performed in patients with stenosis of the vascular access for haemodialysis demonstrated 14% difference in technical success of angioplasty, favouring the 3 minutes balloon inflation time vs one minute. Recently published retrospective single centre study demonstrated that balloon angioplasty with a prolonged inflation time >3 minutes may be effective as an initial angioplasty strategy to prevent severe dissection in femoropopliteal lesions. Type C or higher dissections according to NHLBI (National Heart, Lung and Blood Institute) classification were observed less frequently after >3 minutes balloon inflation - 22.7% vs 50.9% in <3-minute group. However, the rate of provisional stenting was not significantly different between groups.

Objective. The study is aimed to test the hypothesis that a prolonged (6 minutes) time of inflation of angioplasty balloon would reduce the rate of severe (grade C-F) arterial dissections and necessity in bailout stenting during the treatment of occlusive-stenotic femoropopliteal lesions in patients with chronic limb threatening ischemia.

Methods. The LOVES (LOng VErsus Short) trial is a single centre, two parallel groups, open label, controlled trial with 1:1 randomization. The eligible participants in the study will be adults aged 18 years or over who met the inclusion criteria.

Recruitment. Participants in the LOVES trial will be recruited starting with September 2020 among the patients hospitalized in Vascular Surgery Department of Institute of Emergency Medicine, Chisinau, Republic of Moldova. All patients eligible for enrollment in to the study will be asked to sign informed consent. Only one extremity per patient may be included in the trial. If both legs meet the inclusion criteria, the leg with the most severe complaints will be treated first and will be included in the trial.

Procedure. The endovascular intervention will be performed in the dedicated suite under local anesthesia. All types of the arterial access (brachial, femoral crossover, femoral anterograd) will be allowed. After arterial access patients from both arms will receive 5000 IU of heparin intravenously. Diagnostic angiography of the treated limb will be performed first to confirm the presence of stenosis ≥50% or occlusion in the superficial femoral and/or popliteal artery. After successful intraluminal crossing of the femoropopliteal lesion patient will be supposed to randomization.

In the intervention group (long time inflation) the plain old (non drug eluting) angioplasty balloon will be positioned in the affected arterial segment and inflated up to nominal pressure for 6 minutes. In the control group (short time inflation) the plain old (non drug eluting) angioplasty balloon will be positioned in the affected arterial segment and inflated up to nominal pressure for 3 minutes. The length and diameter of the balloon will be selected by operator basing on reference images.

After balloon deflation and extraction the completion angiography will be performed. Presence (yes/no) and severity (grades A-B or C-F according to NHLBI classification) of dissection will be assessed independently by 3 study investigators basing on DSA images in 2 directions. Decision to classify the dissection as severe (grade C-F) and to perform the bailout stenting will be done by the agreement between at least 2 from 3 investigators. Self expandable and balloon expandable non drug eluting stents either will be allowed for implantation.

Additional endovascular interventions in the inflow (aorto-iliac segment) or outflow (infrapopliteal segment) arteries may be performed. These treatments will be registered, reported but not analyzed as study endpoints.

Postoperative antithrombotic treatment will be identical in both groups. After loading dose of clopidogrel (300 mg) patients will receive the 75 mg of clopidogrel and 75 mg of aspirin for 3 months.

Sample size. Basing on the results of previous studies investigators expect the 23% rate of severe dissection in study group (6 minutes inflation) and 51% - in control group (3 minutes inflation). Using the probability of type I error of 0.05 and power set at 80% investigators have calculated that 45 patients are required for each group. Anticipating 10% rate of loss to follow-up, 50 patients will be randomized per treatment arm.

Randomization. Randomization of the patients will be performed by designated study investigator after successful intraluminal crossing of the target lesion. One hundred patients will be allocated to study or control group by two blocks 1:1 randomization using the free online application Research Randomizer, version 4 (http://www.randomizer.org/).

Blinding. Surgeons participating in endovascular procedure and assessing the severity of the dissection can not respect the blinding because their implication in the inflation/deflation of the angioplasty balloon. Patients will be blinded to the treatment they receive. The time of balloon inflation will be not documented in the patient's medical record. Vascular technician who will perform the ABI measurement and duplex ultrasound will be not aware of time of balloon inflation during angioplasty.

Follow-up. Three follow up visits at 1, 6 and 12 months are scheduled according to the standards of management after endovascular peripheral arterial interventions. Physical examination, ABI measurement and duplex ultrasound will be performed during the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic limb threatening ischemia category 4-6 according to Rutherford classification;
2. Ankle-brachial index <0.8 or >1.4
3. Clinical stage ≥2 of WIfI (Wound, Ischemia, foot Infection) classification;
4. Stenosis of ≥50% or occlusion in superficial femoral or popliteal artery, confirmed by duplex ultrasound, computer tomography angiography or digital subtraction angiography;
5. Use of endovascular approach for treatment of the lesion;
6. Patient willing to sign informed consent.

Exclusion Criteria:

1. Acute arterial occlusion (symptoms duration less than 14 days);
2. Recurrent stenosis or occlusion of femoropopliteal segment;
3. Impossibility to cross the lesion intraluminally during the endovascular intervention;
4. Life expectancy of less than 1 year -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Severe post-angioplasty dissection in femoropopliteal arterial segment | 5 minutes after deflation of angioplasty balloon
  Post-angioplasty dissection of grades C-F according to NHLBI (National Heart, Lung and Blood Institute) classification, determined by the agreement between at least 2 from 3 study investigators basing on completion DSA results

SECONDARY OUTCOMES:
Technical success of the procedure | 10 minutes after completion of balloon angioplasty +/- stenting
  Residual stenosis in femoropopliteal segment <30%, according to the DSA
Change in Ankle-Brahial Index | 24 hours after intervention
  Increase or decrease of the ABI by at least 0.1
Primary patency | During the follow-up visits (1, 6, 12 months)
  Absence of occlusion or stenosis ≥50% in femoropopliteal segment assessed by duplex ultrasound (peak systolic velocity ratio >2.5) and freedom from target lesion revascularization
Limb loss | During the follow-up visits (1, 6, 12 months)
  Above the ankle amputation

CONTACTS AND LOCATIONS:
Overall Officials: Dumitru Casian, MD, PhD, Principal Investigator — Nicolae Testemitanu State University of Medicine and Pharmacy
Locations (1):
- Nicolae Testemitanu State University of Medicine and Pharmacy, Department of surgery nr.3, Vascular Surgery Clinic, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zorger N, Manke C, Lenhart M, Finkenzeller T, Djavidani B, Feuerbach S, Link J. Peripheral arterial balloon angioplasty: effect of short versus long balloon inflation times on the morphologic results. J Vasc Interv Radiol. 2002 Apr;13(4):355-9. doi: 10.1016/s1051-0443(07)61736-9. PMID 11932365
- [Background] Forauer AR, Hoffer EK, Homa K. Dialysis access venous stenoses: treatment with balloon angioplasty--1- versus 3-minute inflation times. Radiology. 2008 Oct;249(1):375-81. doi: 10.1148/radiol.2491071845. PMID 18796688
- [Background] Horie K, Tanaka A, Taguri M, Kato S, Inoue N. Impact of Prolonged Inflation Times During Plain Balloon Angioplasty on Angiographic Dissection in Femoropopliteal Lesions. J Endovasc Ther. 2018 Dec;25(6):683-691. doi: 10.1177/1526602818799733. Epub 2018 Sep 11. PMID 30203701